CLINICAL TRIAL: NCT04314167
Title: Effect of Serum LDL Cholesterol Concentration on Pancreatic Insulin Secretion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor recruitment
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 045/2020BO2
Record Dates: First submitted 2020-03-10; First posted 2020-03-19 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Hypercholesterolemia; Insulin Resistance; Insulin Secretion
MeSH Terms: conditions — Hypercholesterolemia; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LDL lowering therapy (Experimental): Patients will receive the PCSK9-inhibitor Evolocumab as part of routine clinical management within the indication of this drug.
  Interventions: Drug: Lowering cholesterol concentrations by PCSK-9 inhibitor

INTERVENTIONS:
Drug: Lowering cholesterol concentrations by PCSK-9 inhibitor — Patients will receive the PCSK9-inhibitor Evolocumab as part of routine clinical management within the indication of this drug.

SUMMARY:
Dyslipidemia is characterized by low levels of HDLs, hypertriglyceridemia as well as an increases proportion of small dense LDLs. Changes in lipoprotein particles and its concentrations, especially increased levels of pro-atherogenic LDL particles play an important role in the development of cardiovascular diseases. It is well established that statin/PCSK9-inhibitor treatment is very effective in lowering LDL cholesterol levels and therefore in preventing cardiovascular events. Besides the beneficial effects on cardiovascular system, these therapies are unfortunately linked to increased risk for type 2 diabetes.

However underlying mechanisms for the association between LDL cholesterol levels and the risk for type 2 diabetes remains largely unknown.Type 2 diabetes is especially characterized by insulin resistance and impaired insulin secretion from pancreatic beta-cells. Insulin resistance alone is insufficient to cause type 2 diabetes, as long as the ß-cell is able to compensate for the increased demand for insulin. Once this compensatory mechanism reaches its physiological limits, individuals progress to type 2 diabetes. Accordingly we aimed to investigate the associations between LDL cholesterol concentrations and the key issue in the pathogenesis of type 2 diabetes, insulin secretion before and after lowering cholesterol concentration by treatment with Evolocumab for 12 weeks in patients with medical indication for a treatment with a PCSK9-inhibitor. Therefore, patients will either undergo a hyperglycemic clamp or a oral glucose tolerance test in randomized manner.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures
* Medical indication for the treatment with a PCSK9-inhibitor
* HbA1c < 6,5%

Exclusion Criteria:

* Diabetes mellitus
* Pregnant women or breastfeeding
* Hb < 11.5 g/dl (males) or Hb < 10.5 g/dl (females)
* treatment with any medication that effects on blood glucose concentrations, e.g. antidiabetic drugs or steroids
* Any pancreatic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Change in insulin secretion. | before and after 12 weeks of treatment with a PCSK9-inhibitor.
  Effect of lowering LDL cholesterol levels on insulins secretion.This will be quantified in half of the patients by a hyperglycemic clamp and in the other half by a 75 g oral glucose tolerance test (randomized assignment).

SECONDARY OUTCOMES:
Change in insulin sensitivity. | before and after 12 weeks of treatment with a PCSK9-inhibitor.
  Effect of lowering LDL cholesterol levels on insulin sensitivity. This will be quantified in half of the patients by a hyperglycemic clamp and in the other half by a 75 g oral glucose tolerance test (randomized assignment).
Change in insulin clearance. | before and after 12 weeks of treatment with a PCSK9-inhibitor.
  Effect of of lowering LDL cholesterol levels on insulin clearance.This will be quantified in half of the patients by a hyperglycemic clamp and in the other half by a 75 g oral glucose tolerance test (randomized assignment).
Change in glucose tolerance. | before and after 12 weeks of treatment with a PCSK9-inhibitor.
  Effect of lowering LDL cholesterol levels on glucose tolerance assessed by 75g oral glucose tolerance test

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tuebingen, Department of Internal Medicine IV, Tübingen, Germany